CLINICAL TRIAL: NCT06144697
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, First-in-human, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Prodrug BMS-986465 and Its Active Derivative, BMS-986464, in Healthy Participants Including Healthy Participants of Japanese Ethnicity and an Open-label Assessment of Food, Formulation, and pH Effects on the Relative Bioavailability of BMS-986465 and BMS-986464
Brief Title: A Study to Evaluate the Safety, Tolerability, Drug Levels, Food, Formulation, and pH Effects on Relative Absorption of BMS-986465 and Its Active Derivative BMS-986464 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN009-1024
Record Dates: First submitted 2023-11-17; First posted 2023-11-22 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants
Keywords: Pharmacokinetics; Pharmacodynamics; Healthy Participants; Healthy Japanese Participants; BMS-986465; SAD; MAD; Safety; Tolerability; Food Effects; Formulation; First-in-human
MeSH Terms: interventions — peginterferon alfa-2a; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Single Ascending Dose (SAD) [BMS-986465 or placebo] (Experimental)
  Interventions: Drug: BMS-986465; Other: Placebo
- Part B: Multiple Ascending Dose (MAD) [BMS-986465 or placebo, Pegasys] (Experimental)
  Interventions: Drug: BMS-986465; Other: Placebo; Drug: Pegasys
- Part C: MAD in Japanese ethnicity [BMS-986465 or placebo] (Experimental)
  Interventions: Drug: BMS-986465; Other: Placebo
- Part D: Food/Formulation/pH Effects [BMS-986465, Famotidine] (Experimental)
  Interventions: Drug: BMS-986465; Drug: Famotidine

INTERVENTIONS:
Drug: BMS-986465 — Specified dose on specified days
Other: Placebo — Specified dose on specified days
  Arms: Part A: Single Ascending Dose (SAD) [BMS-986465 or placebo]; Part B: Multiple Ascending Dose (MAD) [BMS-986465 or placebo, Pegasys]; Part C: MAD in Japanese ethnicity [BMS-986465 or placebo]
Drug: Pegasys — Specified dose on specified days
  Arms: Part B: Multiple Ascending Dose (MAD) [BMS-986465 or placebo, Pegasys]
Drug: Famotidine — Specified dose on specified days
  Arms: Part D: Food/Formulation/pH Effects [BMS-986465, Famotidine]

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, drug and food effects on relative bioavailability of BMS-986465 and its active derivative BMS-986464 in healthy participants and healthy participants of Japanese ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (i e, women not of childbearing potential) participants
* Body Mass Index (BMI) of 18 to 32 kg^m2 and total body weight ≥ 50 kg
* Parts A, B, and D: Participants without restriction on ethnicity
* Part C: Participants of Japanese ethnicity (both biological parents are ethnically Japanese)

Exclusion Criteria:

* Clinically significant medical, psychiatric and/or sound social reason, as determined by the investigator
* Any major surgery within 3 months of study intervention administration
* Participation in another clinical trial concurrent with this study

Note: Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 267 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 28 days
Incidence of serious adverse events (SAEs) | Up to 28 days
Number of participants with vital sign abnormalities | Up to 28 days
Number of participants with physical examination abnormalities | Up to 28 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 28 days
Number of participants with clinical laboratory abnormalities | Up to 28 days
Treatment-emergent suicidal ideation and behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 28 days

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 27
Time of maximum observed plasma concentration (Tmax) | Up to Day 27
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] | Up to Day 27
Cerebrospinal fluid (CSF) concentrations | Up to Day 27
Ratios of CSF to plasma concentrations | Up to 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution - 0001, Anaheim, California
  - Local Institution - 0003, Austin, Texas

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com